CLINICAL TRIAL: NCT06152549
Title: Assessing the Emotional and Physiological Response of Adults to Completing a Self-report Scale on Exposure to Childhood Maltreatment - Online Component
Brief Title: Online Emotional Response to Completing a Childhood Maltreatment Self-report Scale
Acronym: MACEStress
Status: Completed | Type: Observational
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Martin H Teicher, Associate Professor of Psychiatry, Mclean Hospital
Other Study IDs: 401730
Record Dates: First submitted 2022-12-07; First posted 2023-11-30 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Stress, Psychological; Stress, Emotional
Keywords: childhood maltreatment,; adverse childhood experiences; standardized math and verbal tests
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MACE First Group: This group (N=250) will be presented with the Maltreatment and Abuse Chronology of Exposure (MACE) scale toward the beginning of the session and the Math/Verbal Test toward the end.
  Interventions: Behavioral: Maltreatment and Abuse Chronology of Exposure Scale as a stress challenge; Behavioral: Standardized Maths and Verbal Questions such as the ones used in SATs; Behavioral: Chronology of Perceived Discrimination Scale (CPDS); Behavioral: International Personality Item Pool (IPIP-NEO)
- Standardized Test Questions First Group: This group (N=250) will be presented with the standardized test questions (Math/Verbal) toward the beginning of the session and the Maltreatment and Abuse Chronology of Exposure (MACE) scale toward the end.
  Interventions: Behavioral: Maltreatment and Abuse Chronology of Exposure Scale as a stress challenge; Behavioral: Standardized Maths and Verbal Questions such as the ones used in SATs; Behavioral: Chronology of Perceived Discrimination Scale (CPDS); Behavioral: International Personality Item Pool (IPIP-NEO)

INTERVENTIONS:
Behavioral: Maltreatment and Abuse Chronology of Exposure Scale as a stress challenge — The first group (N=250) will receive the Maltreatment and Abuse Chronology of Exposure (MACE) scale first, to assess early life adversity, followed by the standardized test questions. A POMS will be administered before each challenge.
Behavioral: Standardized Maths and Verbal Questions such as the ones used in SATs — The second group (N=250) will be presented with the standardized test questions (Math/Verbal) to assess their stress level, measured through POMS, followed by the Maltreatment and Abuse Chronology of Exposure (MACE) scale.
Behavioral: Chronology of Perceived Discrimination Scale (CPDS) — The group will also receive the Chronology of Perceived Discrimination Scale (CPDS) to assess type and timing of perceived discrimination during the first 18 years of life. A POMS will be administered before and after the intervention/challenge.
Behavioral: International Personality Item Pool (IPIP-NEO) — Participants in both groups will be presented with the abbreviated version of the IPIP-NEO a personality questionnaire that provides ratings on the Five Factor Personality Model. The research team sees this task as non-stressful and even potentially soothing and envisions that it will help to restore an individual's mood before taking the next stressful test and again at the completion of the online session.

SUMMARY:
Childhood adversity in the form of maltreatment and household dysfunction is the most important risk factor for psychopathology as well as a major risk factor for a host of medical disorders. It has been estimated that adverse childhood experiences account for 45%, 50%, 64% and 67% of the population attributable risk for childhood onset psychiatric disorders, alcoholism, depression, substance abuse and suicide attempts. There is also increasing evidence that maltreated and non-maltreated individuals with the same primary psychiatric diagnosis are clinically and neurobiologically distinct and respond differently to treatment. The investigators and others have proposed that assessment of exposure to maltreatment is imperative for prevention, targeted treatment and research. A potential barrier to the widespread collection of data regarding early life stress and childhood maltreatment is the concern that asking such probing questions, particularly on an online questionnaire, may provoke untoward reactions and create clinical problems.

Therefore, the investigators have designed this observational study to test our hypothesis that answering questions about type and timing of childhood maltreatment are no more stressful than answering standardized mathematical and verbal questions, of the type asked on the Scholastic Aptitude Test (SAT).

The study will include representative national samples (by age, sex, and ethnicity) from the United States (total N=500, Ages 18-65) and will be conducted online via Prolific™, which maintains a pool of research participants.

Participants will be assigned randomly to one of two test sequences.

* In sequence 1, the Maltreatment and Abuse Chronology of Exposure (MACE) scale will be presented toward the beginning of the session and the Math/Verbal Test toward the end.
* In sequence 2, the order will be reversed.

The impact of completing the MACE and standardized IQ questions will be assessed before and after each module, using the abbreviated form of the Profile of Mood States (POMS).

DETAILED DESCRIPTION:
Childhood adversity in the form of maltreatment and household dysfunction is the most important risk factor for psychopathology as well as a major risk factor for a host of medical disorders. Briefly, it has been estimated that adverse childhood experiences account for 45%, 50%, 54%, 64% and 67% of the population attributable risk for childhood onset psychiatric disorders, alcoholism, depression, substance abuse and suicide attempts, respectively. Maltreatment is also associated with increased risk for heart disease, cancer, chronic lung disease, liver disease, and shortened life span. There is increasing evidence that maltreated and non-maltreated individuals with the same primary psychiatric diagnosis are clinically and neurobiologically distinct and respond differentially to treatment. Hence, the investigators and others have proposed that assessment of exposure to maltreatment is imperative for prevention, targeted treatment, and research.

However, a potential barrier to widespread collection of data regarding early life stress and childhood maltreatment is the concern that asking such probing questions, particularly on an online questionnaire, may provoke untoward reactions and create clinical problems. To date, the investigators have collected maltreatment data on over 3000 participants without a single call from participants about feeling distressed. While some IRBs permit collection of this information online, the investigators are aware of colleagues at other universities who have had their request denied.

Our thought is that whatever human subjects' limitations should be imposed on collecting childhood maltreatment data via self-report should not simply be a matter of opinion but should be based on evidence.

Hence, the investigators are proposing to specifically study the acute emotional response of volunteer participants, especially those with a history of self-reported childhood maltreatment, to completing a detailed self-report instrument on type and timing of exposure to childhood maltreatment. For contrast, the investigators will also compare their response to completing a series of mathematical and verbal questions, of the type asked on the Scholastic Aptitude Test (SAT), as an example of the type of questions that can be asked without human subject approval.

Our primary hypothesis is that endeavoring to answer these questions will be more stressful and emotionally provocative than questions regarding history of childhood maltreatment, even in participants who report moderate-to-high levels of childhood maltreatment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers ages 18-65, living full-time in the U.S at the time of participation in the study.

Exclusion Criteria:

* Below 18 or above 65. Living outside the U.S at the time of participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Data will be collected online from participants across the USA. The study will include representative national sample (by age, sex, and ethnicity) of healthy volunteers, from the United States (total N=500) and will be conducted via Prolific™, which maintains a pool of research participants specifically interested in participating in online behavioral or psychological research studies.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Profile of Mood States (POMS) | Through study completion, an average of 90 mins
  The abbreviated form of the POMS(40-items) provides ratings of anger-hostility, confusion-bewilderment, depression-dejection, fatigue-inertia, tension-anxiety, vigor-activity, friendliness and a total mood disturbance score. It takes only 3-5 minutes to complete. Items are scored as Not at all(0), A little(1), Moderately(2), Quite a lot(3), Extremely(4). Scores for the seven subscales in the abbreviated POMS are calculated by summing the numerical ratings for items that contribute to each subscale, with two items "Ashamed" and "Embarrassed" reverse scored.
Total Mood Disturbance (TMD) | Through study completion, an average of 90 mins
  Total Mood Disturbance (TMD) is calculated by summing the totals for the POMS negative subscales and then subtracting the totals for the POMS positive subscales.
  The formula is as follows:
  TMD = [Tension+Depression+Anger+Fatigue+Confusion] - [Vigor+Esteem-related Affect]

CONTACTS AND LOCATIONS:
Overall Officials: Martin H Teicher, MD,PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital through ProlificTM, Belmont, Massachusetts, United States

REFERENCES:
- [Background] Anda RF, Brown DW, Dube SR, Bremner JD, Felitti VJ, Giles WH. Adverse childhood experiences and chronic obstructive pulmonary disease in adults. Am J Prev Med. 2008 May;34(5):396-403. doi: 10.1016/j.amepre.2008.02.002. PMID 18407006
- [Background] Anda RF, Whitfield CL, Felitti VJ, Chapman D, Edwards VJ, Dube SR, Williamson DF. Adverse childhood experiences, alcoholic parents, and later risk of alcoholism and depression. Psychiatr Serv. 2002 Aug;53(8):1001-9. doi: 10.1176/appi.ps.53.8.1001. PMID 12161676
- [Background] Brown DW, Anda RF, Felitti VJ, Edwards VJ, Malarcher AM, Croft JB, Giles WH. Adverse childhood experiences are associated with the risk of lung cancer: a prospective cohort study. BMC Public Health. 2010 Jan 19;10:20. doi: 10.1186/1471-2458-10-20. PMID 20085623
- [Background] Brown DW, Anda RF, Tiemeier H, Felitti VJ, Edwards VJ, Croft JB, Giles WH. Adverse childhood experiences and the risk of premature mortality. Am J Prev Med. 2009 Nov;37(5):389-96. doi: 10.1016/j.amepre.2009.06.021. PMID 19840693
- [Background] Dong M, Dube SR, Felitti VJ, Giles WH, Anda RF. Adverse childhood experiences and self-reported liver disease: new insights into the causal pathway. Arch Intern Med. 2003 Sep 8;163(16):1949-56. doi: 10.1001/archinte.163.16.1949. PMID 12963569
- [Background] Dong M, Giles WH, Felitti VJ, Dube SR, Williams JE, Chapman DP, Anda RF. Insights into causal pathways for ischemic heart disease: adverse childhood experiences study. Circulation. 2004 Sep 28;110(13):1761-6. doi: 10.1161/01.CIR.0000143074.54995.7F. Epub 2004 Sep 20. PMID 15381652
- [Background] Dube SR, Anda RF, Felitti VJ, Chapman DP, Williamson DF, Giles WH. Childhood abuse, household dysfunction, and the risk of attempted suicide throughout the life span: findings from the Adverse Childhood Experiences Study. JAMA. 2001 Dec 26;286(24):3089-96. doi: 10.1001/jama.286.24.3089. PMID 11754674
- [Background] Dube SR, Felitti VJ, Dong M, Chapman DP, Giles WH, Anda RF. Childhood abuse, neglect, and household dysfunction and the risk of illicit drug use: the adverse childhood experiences study. Pediatrics. 2003 Mar;111(3):564-72. doi: 10.1542/peds.111.3.564. PMID 12612237
- [Background] Dube SR, Felitti VJ, Dong M, Giles WH, Anda RF. The impact of adverse childhood experiences on health problems: evidence from four birth cohorts dating back to 1900. Prev Med. 2003 Sep;37(3):268-77. doi: 10.1016/s0091-7435(03)00123-3. PMID 12914833
- [Background] Felitti VJ, Anda RF, Nordenberg D, Williamson DF, Spitz AM, Edwards V, Koss MP, Marks JS. Relationship of childhood abuse and household dysfunction to many of the leading causes of death in adults. The Adverse Childhood Experiences (ACE) Study. Am J Prev Med. 1998 May;14(4):245-58. doi: 10.1016/s0749-3797(98)00017-8. PMID 9635069
- [Background] Gordis EB, Granger DA, Susman EJ, Trickett PK. Salivary alpha amylase-cortisol asymmetry in maltreated youth. Horm Behav. 2008 Jan;53(1):96-103. doi: 10.1016/j.yhbeh.2007.09.002. Epub 2007 Sep 12. PMID 17945232
- [Background] Green JG, McLaughlin KA, Berglund PA, Gruber MJ, Sampson NA, Zaslavsky AM, Kessler RC. Childhood adversities and adult psychiatric disorders in the national comorbidity survey replication I: associations with first onset of DSM-IV disorders. Arch Gen Psychiatry. 2010 Feb;67(2):113-23. doi: 10.1001/archgenpsychiatry.2009.186. PMID 20124111
- [Background] Heim C, Newport DJ, Mletzko T, Miller AH, Nemeroff CB. The link between childhood trauma and depression: insights from HPA axis studies in humans. Psychoneuroendocrinology. 2008 Jul;33(6):693-710. doi: 10.1016/j.psyneuen.2008.03.008. PMID 18602762
- [Background] Kirschbaum C, Pirke KM, Hellhammer DH. The 'Trier Social Stress Test'--a tool for investigating psychobiological stress responses in a laboratory setting. Neuropsychobiology. 1993;28(1-2):76-81. doi: 10.1159/000119004. PMID 8255414
- [Background] Monteleone AM, Patriciello G, Ruzzi V, Cimino M, Giorno CD, Steardo L Jr, Monteleone P, Maj M. Deranged emotional and cortisol responses to a psychosocial stressor in anorexia nervosa women with childhood trauma exposure: Evidence for a "maltreated ecophenotype"? J Psychiatr Res. 2018 Sep;104:39-45. doi: 10.1016/j.jpsychires.2018.06.013. Epub 2018 Jun 19. PMID 29936175
- [Background] Navalta CP, Polcari A, Webster DM, Boghossian A, Teicher MH. Effects of childhood sexual abuse on neuropsychological and cognitive function in college women. J Neuropsychiatry Clin Neurosci. 2006 Winter;18(1):45-53. doi: 10.1176/jnp.18.1.45. PMID 16525070
- [Background] Nemeroff CB, Heim CM, Thase ME, Klein DN, Rush AJ, Schatzberg AF, Ninan PT, McCullough JP Jr, Weiss PM, Dunner DL, Rothbaum BO, Kornstein S, Keitner G, Keller MB. Differential responses to psychotherapy versus pharmacotherapy in patients with chronic forms of major depression and childhood trauma. Proc Natl Acad Sci U S A. 2003 Nov 25;100(24):14293-6. doi: 10.1073/pnas.2336126100. Epub 2003 Nov 13. PMID 14615578
- [Background] Obayashi K. Salivary mental stress proteins. Clin Chim Acta. 2013 Oct 21;425:196-201. doi: 10.1016/j.cca.2013.07.028. Epub 2013 Aug 9. PMID 23939251
- [Background] Teicher MH, Samson JA. Childhood maltreatment and psychopathology: A case for ecophenotypic variants as clinically and neurobiologically distinct subtypes. Am J Psychiatry. 2013 Oct;170(10):1114-33. doi: 10.1176/appi.ajp.2013.12070957. PMID 23982148
- [Background] Williams LM, Debattista C, Duchemin AM, Schatzberg AF, Nemeroff CB. Childhood trauma predicts antidepressant response in adults with major depression: data from the randomized international study to predict optimized treatment for depression. Transl Psychiatry. 2016 May 3;6(5):e799. doi: 10.1038/tp.2016.61. PMID 27138798
- [Result] Grove, J.R., & Prapavessis, H. (1992). Preliminary evidence for the reliability and validity of an abbreviated Profile of Mood States. International Journal of Sport Psychology, 23, 93-109.
- [Result] Norcross JC, Guadagnoli E, Prochaska JO. Factor structure of the Profile of Mood States (POMS): two partial replications. J Clin Psychol. 1984 Sep;40(5):1270-7. doi: 10.1002/1097-4679(198409)40:53.0.co;2-7. PMID 6490926
- [Result] Shichiri, K. , Shibuya, M. , Watanabe, M. , Tahashi, M. , Kaminushi, K. , Uenoyama, T. , Mashima, I. , Murayama, K. , Kuroda, T. and Suzuki, Y. (2016) Correlations between the Profile of Mood States (POMS) and the WHOQOL-26 among Japanese University Students. Health, 8, 416-420. doi: 10.4236/health.2016.85044.